CLINICAL TRIAL: NCT02309580
Title: A Multicenter Phase I Study of Ibrutinib in Relapsed and Refractory T-cell Lymphoma
Brief Title: Study of Ibrutinib in Relapsed and Refractory T-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Ohio State University (Other); Pharmacyclics LLC. (Industry); Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-227
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: T-cell Lymphoma; Relapsed and Refractory T-cell Lymphoma
Keywords: Ibrutinib; 14-227
MeSH Terms: conditions — Lymphoma, T-Cell; Recurrence | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ibrutinib (Experimental): This will be a standard dose-escalation study to determine the MTD of ibrutinib in relapsed/refractory PTCL or CTCL. At each dose 6 patients with TCL (PTCL or CTCL) will be enrolled. The first 6 patients will be enrolled at dose level 1. Dose escalation to the next dose level will proceed after DLT assessment of all 6 patients at the end of cycle 1 (28-days).
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib will be administered once daily continuously until disease progression (confirmed by two assessments for CTCL patients only) or intolerance. The dose levels for the Phase 1 portion of the study. Either 560 mg (4 X 140 mg capsules) or 840 mg (6 X 140 mg capsules) doses will be administered. After the recommended expansion dose is established, an expansion cohort of 12 additional patients will be treated at the recommended expansion dose to further characterize the safety at that dose and to further assess preliminary efficacy

SUMMARY:
This is a Phase 1 clinical trial, a type of research study. The purpose of this phase 1 clinical trial is to find out whether a new study drug, ibrutinib, is safe in patients with T-cell non-Hodgkin lymphoma that has either come back or not responded to treatment. In this phase 1 study, different doses of ibrutinib (560 mg and 840 mg daily) will be tested to see what effect the drug has on the patient and the disease.

ELIGIBILITY:
Inclusion Criteria:

* Pathology confirmed relapsed or refractory T-cell lymphoma (PTCL and stage >IBCTCL) at treating institution
* Relapse or progression after at least 1 systemic therapy
* Age ≥18 years at the time of signing the informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Previous systemic anti-cancer therapy must have been discontinued at least 3 weeks prior to treatment in this study. If there is progression of disease on that therapy and all adverse effects have resolved to Grade 1 or baseline, in which case 2 weeks is acceptable
* Previous radiation, hormonal therapy, and surgery must have been discontinued at least 2 weeks prior to treatment in this study and adverse effects must have resolved. Lymph node or other diagnostic biopsy within 2 weeks is not considered exclusionary
* Systemic corticosteroids are permissible in the following circumstances:
* Short course systemic corticosteroids for disease control, improvement of performance status or non-cancer indication (≤ 7 days) must have been discontinued at least 7 days prior to study treatment.
* Ongoing administration of a stable dose of corticosteroid therapy (previously received for ≥ 30 days) is permissible provided there is evidence of measurable disease and there will be no increase in steroid dose during the clinical trial
* ECOG performance status of ≤ 2 at study entry
* Patients who have undergone autologous stem cell transplant > 6 months prior are eligible
* Patients who have undergone allogeneic stem cell transplant > 12 months, without active graft-versus-host-disease, and not on immunosuppression for prevention of graft-versus-host disease are eligible
* Laboratory test results within these range:
* Adequate hematologic function with screening laboratory assessment defined as:
* Absolute neutrophil count >1,000 cells/mm3 (1.0 x 10^9/L)
* Platelet count >75,000 cells/mm3 (75 x 10^9/L), if thrombocytopenia is due to bone marrow involvement platelet count must be ≥ 50,000 cells/mm3
* Hemoglobin >8.0 g/dL
* Adequate hepatic and renal function with screening laboratory assessment defined as:
* Serum aspartate transaminase (AST) or alanine transaminase (ALT)

  ≤2.5 x upper limit of normal (ULN)
* Creatinine <2.0 x ULN or Estimated Glomerular Filtration Rate GFR [Cockcroft-Gault] > 30 mL/min.
* Bilirubin <1.5 x ULN [unless bilirubin rise is due to Gilbert's syndrome (as defined by >80% unconjugated hyperbilirubinemia) or of nonhepatic origin]
* Females of childbearing potential (FCBP)† must have a negative serum pregnancy test and agree to use appropriate methods of birth control

Exclusion Criteria:

* Patients who have a standard curative option for their lymphoid malignancy at current state of disease are excluded. For eligibility on this trial, allogeneic stem cell transplantation is not considered a standard curative option
* Concurrent systemic immunosuppressant therapy (eg, cyclosporine A, tacrolimus, etc.) within 28 days of the first dose of study drug
* Recent infection requiring intravenous anti-infective treatment that was completed ≤14 days before the first dose of study drug
* Known bleeding diathesis (eg, von Willebrand's disease) or hemophilia
* Treatment with warfarin or other Vitamin K antagonists (eg, phenprocoumon)
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the opinion of the investigator, could compromise the subject's safety or put the study outcomes at undue risk
* Unwilling or unable to participate in all required study evaluations and procedures.
* Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF)
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to enrollment
* Unable to swallow capsules, malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction
* Pregnant females (Lactating females must agree not to breast feed while taking ibrutinib
* Prior use of ibrutinib
* Known seropositive and requiring anti-viral therapy for human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) defined by PCR.
* Active concurrent malignancy requiring active therapy
* Known central nervous system or meningeal involvement (in the absence of symptoms investigation into central nervous system involvement is not required)
* Patients who require treatment with a strong cytochrome P450 (CYP) 3A inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-01; Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated does | 1 year
  evaluate the safety and toxicities of ibrutinib in patients with relapsed/refractory Tcell lymphoma (PTCL and CTCL) as defined by CTCAE version 4.

SECONDARY OUTCOMES:
overall response rate (ORR) | 1 year
  Response and progression of disease will be evaluated in this study using the revised response criteria for malignant lymphoma with incorporation of PET/CT.33 Response in subjects with CTCL will be assessed using a specific skin scoring system with mSWAT and incorporation of measurements of extracutaneous disease.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Kumar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University, Columbus, Ohio

REFERENCES:
- [Derived] Kumar A, Vardhana S, Moskowitz AJ, Porcu P, Dogan A, Dubovsky JA, Matasar MJ, Zhang Z, Younes A, Horwitz SM. Pilot trial of ibrutinib in patients with relapsed or refractory T-cell lymphoma. Blood Adv. 2018 Apr 24;2(8):871-876. doi: 10.1182/bloodadvances.2017011916. PMID 29669753
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/